CLINICAL TRIAL: NCT04664803
Title: A Clinical Trial to Re-confirm the Efficacy and the Safety of Cefetamet Pivoxil Formulation in Sinusitis Patients: Double Blinded, Randomized, Parallel Designed, Multi-center, Active Comparator Study (CASIS Study)
Brief Title: Safety and Efficacy of Cefecin Tab. in Patients With Acute Sinusitis
Acronym: CASIS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Korea United Pharm. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUP-CFC-401
Record Dates: First submitted 2020-11-24; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-11

CONDITIONS: Acute Sinusitis
MeSH Terms: interventions — cefetamet pivoxyl; Cefdinir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Device: No

ARMS (2):
- Cefecin Tab. (Experimental): Cefecin Tab./Placebo to Omnicef Cap.
  Interventions: Drug: Cefecin Tab.
- Omnicef Cap. (Active Comparator): Omnicef Cap./Placebo to Cefecin Tab.
  Interventions: Drug: Omnicef Cap.

INTERVENTIONS:
Drug: Cefecin Tab.
  Other Names: cefetamet pivoxil
  Arms: Cefecin Tab.
Drug: Omnicef Cap.
  Other Names: cefdinir
  Arms: Omnicef Cap.

SUMMARY:
This is a multi-center, double-blind, randomized, active controlled, parallel group phase 4 clinical trial to re-confirm the efficacy and safety of cefetamet pivoxil formulation in sinusitis patients

DETAILED DESCRIPTION:
Patients with acute sinusitis were randomly assigned (1:1) to receive either cefetamet (500 mg twice daily, study group) or cefdinir (100 mg three times a day, control group) and corresponding placebo t.i.d. or b.i.d. for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with sinusitis (accompanied with otitis media) at screening, and whose first symptoms occurred within the past 3 weeks
* Symptoms or signs of acute sinusitis persist without improvement for 10 days after onset or symptoms or signs of acute sinusitis initially improve and then worsen within 10 days

Exclusion Criteria:

* Those who have a history of hypersensitivity to cephalosporin, penicillin, or other beta-lactam antibiotics
* Those with a history of allergic rhinitis or other rhinitis
* Those who have been diagnosed with sinusitis more than 3 times within a year
* Have had or scheduled sinus surgery within 1 month
* Creatinine Clearance < 40 mL/min at screening
* Those whose AST, ALT, and total bilirubin are more than 3 times the upper limit of normal at screening
* Cystic fibrosis patients

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical effective rate | 21 days
  Percentage of patients with clinical cure and improvement on days 14 and 21

SECONDARY OUTCOMES:
Clinical cure rate | 21 days
  Percentage of patients with clinical cure on days 14 and 21
Clinical effective rate | 14 days
  Percentage of patients with clinical cure and improvement on days 14
Change from baseline in total score of clinical signs | 14 days
  Evaluation of clinical signs through nasal endoscopy; purulent secretion from sinus ostia, pain over sinuses, facial swelling
Change from baseline in total score of clinical signs | 21 days
  Evaluation of clinical signs through nasal endoscopy; purulent secretion from sinus ostia, pain over sinuses, facial swelling